CLINICAL TRIAL: NCT02353650
Title: The Effect of Coenzyme Q10 on Hearing and Tinnitus Characteristics of Chronic Tinnitus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZA, Ethics Committee, University Hospital, Antwerp
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14/27/286
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Tinnitus
Keywords: Q10; ubiquinol
MeSH Terms: conditions — Tinnitus | interventions — Tuberculin; ubiquinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Dietary Supplement: Q10
  Other Names: Ubiquinol
Dietary Supplement: placebo

SUMMARY:
The study is a randomised double-blinded trial. A group of 40 tinnitus patients with a naturally low Q10 level will be selected out of a preselected group of 160 screened out of a pre-existed database or patients which visited the ENT-consultation. The 40 patients with the lowest level will be asked to take 2 months Q10 (n=20) or the placebo (n=20). To evaluate the effect on hearing and tinnitus characteristic; audiometric test, tinnitus analysis and auditory evoked responses will be used as outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* chronic non-pulsatile tinnitus > 3 months
* tinnitus has a clear otological cause
* age > 18 years

Exclusion Criteria:

* pulsatile tinnitus
* persons who take already Q10
* pregnancy
* cervical tinnitus
* holocranial tinnitus
* depression
* mental of neurological disorders
* history of chemotherapy
* middle ear diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-11; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index | 2 months

SECONDARY OUTCOMES:
Audiometric tresholds test | 2 months
Tinnitus Analysis _ loudness matches | 2 months
Tinnitus Analysis_Minimal masking level | 2 months
Visual Analogue Scale of loudness | 2 months
Hospital Anxiety and Depression Scale | 2 months
Hyperacusis Questionnaire | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Antwerp, Edegem, Antwerp, Belgium